CLINICAL TRIAL: NCT05953493
Title: Evaluation of Oxygen Reserve Index According to Glasgow Coma Scale in Providing Oxygenation in Intracranial Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ars Gor Dr Burak Akpinar, Research Assistant Doctor, Trakya University
Other Study IDs: Trakya University
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Oxygen Reserve Index Values

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GKS1: Patients with a Glasgow coma scale between 9 and 12
- GKS2: Patients with a Glasgow coma scale between 13 and 15

SUMMARY:
Evaluation of oxygen reserve index according to Glasgow Coma Scale in providing oxygenation in intracranial surgery

DETAILED DESCRIPTION:
Peroperative oxygenation is one of the most important parameters in providing cerebral blood flow in intracranial surgeries. SpO2, which is included in standard monitoring, is used to show perioperative hypoxia. Although blood gas analysis used in the evaluation of hypoxia is the gold standard for measurement of oxygenation, it is invasive and impractical. For these reasons, oxygen reserve index (ORI) monitoring, which can detect hypoxia earlier than Spo2 measurement and does not require invasive procedures, is a valuable parameter. Patients with different Glasgow Coma Scale (GCS) values may also have different susceptibility to hypoxia. This study aims to evaluate the effectiveness of ORI monitoring in detecting hypoxia and its correlation with SPO2 in providing oxygenation in patients with different GCS values in intracranial surgery.

Method: 150 patients in the ASA I-II-III risk group between the ages of 18-80 who will undergo intracranial surgery by Brain and Nerve Surgery at Trakya University Medical Faculty Hospital will be included in the study. Patients who cannot insert a sensor due to finger deformity or hypoperfusion, intubation difficulty, who have cardiac or pulmonary disease, and preoperative anemia due to hemoglobinopathies will be excluded from the study. When the patients are taken to the operating table, they will be monitored and the input values will be recorded, and they will be divided into two different patient groups as GCS values (9-12) and (13-15). During intracranial surgery; ORI, blood gas, and SPO2 measurements will be recorded during baseline, induction, intubation, pin application, skin incision, craniotomy, dural opening, aneurysm clipping, bleeding control, pin removal, and skin closure. All hemodynamic parameters of the patients such as blood pressure, heart rate, SpO2, ORI, BIS (Bispectral index) values, oxygen saturation, Et CO2, SpO2;% during anesthesia, operation type, operation time, amounts of used anesthetic and analgesic agents, from anesthesia document, will be saved from files and monitors. Postoperative recovery scores (Modified Alderate scoring), VAS values on the first day (1, 2, 4, 6, 12, 24 hours) and analgesics used, time of first postoperative analgesia use and developing complications will be recorded.

Statistics: The suitability of the data to the normal distribution will be examined with the one-sample Kolmogorov Smirnov Test. Student's t-test will be used to compare the quantitative values with normal distribution between the groups, and the Mann-Whitney U test will be used to compare those that do not show normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* 150 patients in the ASA I-II-III risk group between the ages of 18-80 who will undergo intracranial surgery by Brain and Nerve Surgery at Trakya University Medical Faculty Hospital will be included in the study

Exclusion Criteria:

* Patients who cannot insert a sensor due to finger deformity or hypoperfusion, intubation difficulty, who have cardiac or pulmonary disease, and preoperative anemia due to hemoglobinopathies will be excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: intracranial surgery patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
ORI values | March 1, 2022-October 1, 2024
  Comparison of ori values according to the glaskow coma scale

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya Universiy, Edirne, Turkey (Türkiye)